CLINICAL TRIAL: NCT01955785
Title: Respiratory Treatment of Patients With Moderate and Severe Traumatic Brain Injury: A Randomised Comparison of Pressure Controlled Ventilation and Pressure Regulated Volume Controlled Ventilation
Brief Title: Respiratory Treatment of Patients With Moderate and Severe Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/1346
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; Intracranial pressure; Ventilation; Respiratory therapy
MeSH Terms: conditions — Brain Injuries, Traumatic; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PC ventilation (Active Comparator): Intervention with pressure controlled ventilator
  Interventions: Device: pressure controlled ventilator
- PRVC ventilation (Active Comparator): Intervention with Pressure Regulated Volume Controlled Ventilator
  Interventions: Device: Pressure Regulated Volume Controlled Ventilator

INTERVENTIONS:
Device: pressure controlled ventilator
  Arms: PC ventilation
Device: Pressure Regulated Volume Controlled Ventilator
  Arms: PRVC ventilation

SUMMARY:
Intracranial pressure (ICP) in patients with traumatic brain injury (TBI) is influenced by several factors of which one is arterial CO2 tension. Patient with TBI are often sedated and mechanically ventilated in order to secure a stable PaCO2. This study compares two ventilation modus; Pressure Controlled Ventilation (PC) and Pressure Regulated Volume Controlled ventilation (PRVC) in order to observe which of the two ventilation strategies results in a more stable ICP and arterial CO2 pressure (PaCO2).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from the patients next-of-kin.
* moderate or severe TBI according to Head Injury Severity Scale (Glasgow Coma Scale (GCS) score 3-13).
* treated at the neurosurgical ICU or the main ICU at St Olav University Hospital.
* intubated and receiving controlled mechanical ventilation.
* continuous measurement of ICP with either an intraventricular or an intraparenchymal pressure monitor device.
* sedation to a level of sedation corresponding to MAAS (Motor Activity Assessment Score) 0 or 1 with continuous intravenous infusions of midazolam/propofol and morphine/fentanyl/remifentanil14.

Exclusion Criteria:

* Pregnancy
* ICP above 25 mmHg
* ongoing cerebral anti edema therapy corresponding to Step III at St Olav University Hospital therapy guideline
* continuous external drainage of cerebrospinal fluid (CSF)
* Clinical pulmonary condition prohibiting changes in respiratory therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
ICP | Two hours
  Each study period is two hours. All patients receive several study periods (max number 6) in a N=1 design

SECONDARY OUTCOMES:
PaCO2 | Two hours
  Each subject is studied in several study periods each of two hours duration (max number 6 periods). N=1 design

CONTACTS AND LOCATIONS:
Overall Officials: Pål Klepstad, MD PhD, Principal Investigator — National Taiwan Normal University
Locations (1):
- Dept Intensive Care Medicine, St Olavs University Hospital, Trondheim, Norway

REFERENCES:
- [Result] Schirmer-Mikalsen K, Vik A, Skogvoll E, Moen KG, Solheim O, Klepstad P. Intracranial Pressure During Pressure Control and Pressure-Regulated Volume Control Ventilation in Patients with Traumatic Brain Injury: A Randomized Crossover trial. Neurocrit Care. 2016 Jun;24(3):332-41. doi: 10.1007/s12028-015-0208-8. PMID 26503512